CLINICAL TRIAL: NCT05709496
Title: A Feasibility Study of Dose De-escalation in Prostate Radiotherapy Using the Magnetic Resonance Linear Accelerator (MRL)
Brief Title: Dose De-escalation in Prostate Radiotherapy Using the MRL
Acronym: DESTINATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR5715
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Prostate Adenocarcinoma
Keywords: Intermediate risk

STUDY DESIGN:
Intervention Model Description: An R-IDEAL stage 2a study aiming to demonstrate technical feasibility and establish likely toxicity rates for powering the subsequent study.
  Men will receive de-escalated radiotherapy to the prostate with a boost to the dominant lesion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- De-escalated radiotherapy to the prostate (Experimental): De-escalated radiotherapy to the prostate with an intra-prostatic boost to the dominant .
  Interventions: Radiation: De-escalated radiotherapy to be delivered on the Elekta Unity Unity MR-linac

INTERVENTIONS:
Radiation: De-escalated radiotherapy to be delivered on the Elekta Unity Unity MR-linac — 30 Gy in 5 fractions to the whole prostate with 45 Gy in 5 fractions to the dominant lesion

SUMMARY:
The goal of this feasibility study is to learn about dose de-escalation in the treatment of men with intermediate risk prostate cancer.

The main question it aims to answer is the technical feasibility of treating prostate cancer with toxicity-minimising radiotherapy on an Magnetic Resonance Linear Accelerator (MR-linac). It will also examine gastrointestinal and genitourinary toxicity in the acute and late setting post radiotherapy as well as Prostate-Specific antigen (PSA) control up until 2 years post treatment.

Participants will be treated with radiotherapy to the prostate with which will be given in 30Gy in 5 fractions to the whole prostate and 45Gy in 5 fractions to the dominant lesion.

DETAILED DESCRIPTION:
DESTINATION is a single centre phase II non-randomised study in men with intermediate risk localised prostate cancer.

The aim is to establish the technical feasibility of treating prostate cancer with toxicity-minimising radiotherapy on an MR-linac.

20 men will be recruited to take part. All radiotherapy will be delivered on the MR-linac. The whole prostate with no margin will be treated to 30 Gray (Gy) in 5 fractions (i.e. dose to 95% of the Clinical Target Volume prostate should receive 30 Gy (D95%CTVp= 30 Gy)). The dominant lesion (Gross tumour volume (GTV)) as defined on pre-biopsy multiparametric magnetic resonance imaging (mpMRI) plus a 4mm intra-prostatic margin (GTV4mm) will be treated to 45 Gy in 5 fractions, providing standard organ at risk (OAR) constraints can be met. If not, then dose coverage of the GTV will be reduced until the OAR constraints are met (i.e. isotoxic dose escalation). OAR constraints will be as per international standard levels, and largely consistent with the PACE B trial.

The primary end point will be assessed once 14 patients have completed their radiotherapy treatment on the MR-Linac. If any of the first 14 patients do not complete all five fractions planned, then recruitment will continue until we have 14 assessable patients. The analysis population for the primary endpoint will be defined as those patients who have completed all five fractions of stereotactic body radiotherapy (SBRT) as intended.

If shown to be feasible a total of 20 patients will be recruited to enable a better estimation of the toxicity rates and to further technical proficiency with this technique.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥18 years
* Histological confirmation of prostate adenocarcinoma requiring radical radiotherapy
* Gleason score 3+3, 3+4 or 4+3 (Grade groups 1, 2 or 3)
* MRI stage T2 or less (as staged by AJCC TNM 2018)
* MRI-visible tumour(s) of Prostate Imaging-Reporting and Data System (PIRADS) v2 grade 3 or higher on T2 and diffusion-weighted imaging and/or dynamic contrast-enhanced imaging with concordant pathology
* Tumour nodule visible on MRI occupying <50% of prostate on any axial slice and <50% total prostate volume
* PSA <20 ng/ml prior to starting androgen deprivation therapy (ADT)
* Patients can be concurrently treated with androgen deprivation therapy if this would be standard of care. Luteinizing hormone-releasing hormone (LHRH) analogues or Bicalutamide are permitted. ADT is not mandatory where this would usually be omitted.
* World Health Organisation (WHO) Performance status 0-2
* Ability of the participant understand and the willingness to sign a written informed consent form.
* Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

* Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
* IPSS 19 or higher
* High grade disease (GG3) occult to MRI-defined lesion
* Post-void residual >100 mls, where known
* Prostate volume >90cc
* Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
* Unilateral or bilateral total hip replacement, or other pelvic metalwork which causes artefact on diffusion-weighted imaging
* Previous pelvic radiotherapy
* Patients needing >6 months of ADT due to disease parameters.
* Previous invasive malignancy within the last 2 years excluding basal or squamous cell carcinomas of the skin, low risk non-muscle invasive bladder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a feasibility study in men with intermediate risk prostate cancer
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The technical ability to treat prostate cancer with escalated dose to the gross tumour volume tumour and de-escalated dose to the normal prostate the Unity MR-linac. | 2 years
  The primary end point is defined by coverage of GTV4mm D90% >42Gy on the post-treatment imaging.

SECONDARY OUTCOMES:
Acute toxicity | 2 years
  Physician reported genitourinary (GU) and gastrointestinal (GI) toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) to be taken at baseline and the end of treatment then at 4 and 12 weeks post-treatment.
  The higher the grade the worse the toxicity reported. Each domain will be scored individually.
Late toxicity | 2 years
  Physician reported GU and gastrointestinal (GI) late toxicity (CTCAE) at 1 and 2 years post-treatment.
  The CTCAE toxicity will be graded by the physician, with the higher scores equating to worse toxicity. Each domain will be scored individually.
Patient-reported outcomes | 2 years
  Patient-reported outcome measures (PROMs) from the Expanded Prostate Cancer Index Composite-26 (EPIC-26), (International prostate symptom score) IPSS, and International Index of Erectile Function-5 (IIEF-5) questionnaires. Patients will be asked to complete these PROMs at 4 and 12 weeks, 6 months, 1 and 2 years post treatment.
  EPIC-26 is scored out of 100, with 100 being the best score. IPPS is made of seven questions with lower scores equating to fewer symptoms. IIEF-5 is composed of 5 questions, the highest score of 25 is indicative of severe erectile dysfunction
Biochemical control | 2 years
  The trend in PSA will be measured up until two years. An increase in the PSA is suggested of biochemical failure and disease relapse

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
It is intended that data will be shared within the MOMENTUM collaboration, between centres delivering treatment in the same way as DESTINATION. Pseudonymised data will storage with in MOMENTUM for at least 5 years. Storage will be cloud based and as the treating centre we will have free access to the data and control over who else can assess it.
Supporting Information: Study Protocol, CSR
Time Frame: 5 years
Access Criteria: Must have approved access from the site sponsor.